CLINICAL TRIAL: NCT00596843
Title: Chronic Hepatitis Intervention Project for Drug Users
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DESPR DA013763; R01DA013763-01A2 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-17 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2008-11

CONDITIONS: HIV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Motivational Interviewing; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Motivational intervention
  Interventions: Behavioral: Motivational interviewing
- 2 (Active Comparator): Educational intervention
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Motivational interviewing — 6 one-on-one individual sessions lasting from 30 minutes to 1-hour each
  Arms: 1
Behavioral: Educational intervention — 6 1-hour sessions. 2 sessions are delivered by an interventionist and 4 sessions are delivered as videos
  Arms: 2

SUMMARY:
The purpose of this study is to determine if a 6-session motivational interviewing intervention is more effective than a 6-session educational intervention at reducing behaviors that may lead to infection, transmission, and progression of HIV and hepatitis C among out of treatment injecting drug users.

DETAILED DESCRIPTION:
This 4.5-year community-based study is a randomized field experiment that uses a two-group design. Participants are randomized into either an Educational intervention group or a Motivational intervention group. We are comparing the effectiveness of the Motivational intervention with the Educational intervention. We are also estimating the costs and evaluating the cost-effectiveness of the Motivational intervention relative to the Educational intervention.

We have the following aims and related hypotheses:

Aim 1: To compare the effectiveness of a 6-session personalized motivational intervention to a 6-session educational intervention in terms of injection risk, sexual behavior, alcohol use, and knowledge and perception related to HBV and HCV; H1. Relative to the Educational intervention group, a greater proportion of the Motivational intervention group will report no injection risk at 6- and 12-month follow-up interviews. No injection risk is operationally defined as either no injections in the past 30 days, or no direct or indirect sharing of syringes and other injection equipment in the past 30 days.

H2. Relative to the Educational intervention group, a greater proportion of the Motivational intervention group will report no sexual risk at 6- and 12-month follow-up interviews. No sexual risk is operationally defined as either no sex (oral, vaginal, or anal) in the past 30 days, or no unprotected oral, vaginal, or anal sex in the past 30 days.

H3. Relative to the Educational intervention group, the Motivational intervention group will report greater decreases in frequency of alcohol consumption and quantity of alcohol consumed. Frequency of alcohol consumption is defined as "number of days drank alcohol in the past 30 days," and quantity of alcohol consumed is defined as "the average number of drinks per drinking day during the past 30 days." H4. Relative to the Educational intervention group, participants in the Motivational intervention group will report greater increases in knowledge and more accurate perceptions of severity of disease and efficacy of protective actions regarding hepatitis B and C at Session 3.

Aim 2: To estimate the cost and cost-effectiveness of a 6-session personalized motivational intervention relative to a 6-session educational intervention.

H5. The Motivational Intervention will cost more than the Educational Intervention, but will be cost-effective at eliminating injection risk behavior and sexual risk behavior and at reducing alcohol use

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years injected illicit drugs within last 30 days

Exclusion Criteria:

* participated in formal substance treatment in last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2003-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Reduction/cessation of alcohol use | 6-months and 12-months

SECONDARY OUTCOMES:
Reductions in direct and indirect needle and syringe sharing | 6-months and 12-months
Reductions in unprotected sexual behavior | 6-months and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: William A. Zule, Dr.P.H., Principal Investigator — RTI International
Locations (1):
- RTI International Field Site, Durham, North Carolina, United States

REFERENCES:
- [Result] Zule WA, Costenbader EC, Coomes CM, Wechsberg WM. Effects of a hepatitis C virus educational intervention or a motivational intervention on alcohol use, injection drug use, and sexual risk behaviors among injection drug users. Am J Public Health. 2009 Apr;99 Suppl 1(Suppl 1):S180-6. doi: 10.2105/AJPH.2007.126854. Epub 2009 Feb 12. PMID 19218179